CLINICAL TRIAL: NCT01630824
Title: Development an Effects of a Structural Education Programm in Adult Kidney Transplant Recipients
Brief Title: Development and Effects of a Structural Education Program in Adult Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jena (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Claudia Schinkoethe, Dr. med. Claudia Schinkoethe, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NTXEdu2012
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Kidney Disease
Keywords: education program; kidney transplantation; renal transplantation; evaluation
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Other): Kidney transplant recipients, who undergo the structured education program
  Interventions: Other: Structured education program
- Control (No Intervention): Kidney transplant recipients without structured education programm

INTERVENTIONS:
Other: Structured education program — structured education program after kidney transplantation
  Arms: Education

SUMMARY:
Kidney transplantation is the treatment of choice for patients with end-stage renal disease. The purpose of this randomized and controlled study is to evaluate the efficacy of a structured education program for adult kidney transplant recipients. Patients are randomly assigned to an educational program or to a standard care control group. The education group receives 8 lessons (each 90 minutes, 1 lesson per day), starting 4 days after kidney transplantation. Kidney transplant survival, number of rejections, infectious complications, length of hospital stay, blood pressure, HbA1c, glomerular filtration rate, quality of life (QoL) and knowledge are measured in both groups after 6, 12 and 24 months. The investigators postulate that the education group will have superior outcomes compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years recently had a kidney transplantation able to speak, write and understand german willing to participate regular visits after kidney transplantation

Exclusion Criteria:

* severe complications after recent kidney transplantation early loss of the kidney allograft severe allograft dysfunction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
transplant survival | 2 years

SECONDARY OUTCOMES:
number of rejections | 2 years
days at hospital | 2 years
blood pressure control | 2 years
number of infectious complications | 2 years
quality of life (QoL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gunter Wolf, Principal Investigator — University of Jena
Locations (1):
- Department of Nephrology, University of Jena, Jena, Thuringia, Germany